CLINICAL TRIAL: NCT01328470
Title: Platelet Reactivity in Patients With Chronic Kidney Disease Receiving Adjunctive Cilostazol Compared to a High-maintenance Dose of Clopidogrel
Brief Title: Effect of Platelet Inhibition According to Clopidogrel Dose in Patients With Chronic Kidney Disease
Acronym: CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Kyunghee University, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIANO-CKD2
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Disease; Stable Angina
Keywords: platelet; cilostazol; clopidogrel; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Angina, Stable | interventions — Clopidogrel; Cilostazol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- clopidogrel 75 mg/day (Active Comparator): CKD patients undergoing chronic hemodialysis and PCI for stable coronary artery disease will be randomized to receive clopidogrel 75 mg/day for 14 days.
  Interventions: Drug: Clopidogrel, cilostazol
- clopidogrel 150 mg/day (Active Comparator): CKD patients undergoing chronic hemodialysis and PCI for stable coronary artery disease will be randomized to receive clopidogrel 150 mg/day for 14 days.
  Interventions: Drug: Clopidogrel, cilostazol
- adjunctive cilostazol (Active Comparator): CKD patients undergoing chronic hemodialysis and PCI for stable coronary artery disease will be randomized to receive co-administration of adjunctive cilostazol (100 mg twice daily) and clopidogrel (75 mg/day; [group 3, 20 patients]) for 14 days.
  Interventions: Drug: Clopidogrel, cilostazol
- 75mg clopidogrel (Active Comparator): control group undergoing PCI for stable angina will be also maintained on clopidogrel (75 mg/day for 14 days).
  Interventions: Drug: Clopidogrel, cilostazol

INTERVENTIONS:
Drug: Clopidogrel, cilostazol — Patients with CKD received clopidogrel (75 mg/day)for 14 days Patients with CKD received clopidogrel (150 mg/day)for 14 days Patients with CKD received clopidogrel (75 mg/day)and cilostazol (100 mg twice daily)for 14 days 75mg clopidogrel in patients with normal kidney function for 14 days
  Other Names: Plavix; pletaal

SUMMARY:
Impaired renal function is associated with reduced responsiveness to clopidogrel. There are no studies which have shown a means by which to overcome platelet hyporesponsiveness in patients with chronic kidney disease (CKD). The purpose of this study was to determine the functional impact of cilostazol in patients with CKD undergoing hemodialysis.

DETAILED DESCRIPTION:
The aims of this study is to evaluate the effects of platelet responsiveness to clopidogrel or cilostazol in CKD patients undergoing hemodialysis. The differences in platelet activation markers are also evaluated before and after clopidogrel or cilostazol administration. The investigators will perform a prospective, randomized study to compare the degree of platelet inhibition and platelet activation markers by adjunctive cilostazol (100 mg twice daily) compared to clopidogrel (75 or 150 mg/day) in CKD patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients undergoing chronic hemodialysis and PCI for stable coronary artery disease

Exclusion Criteria:

* known allergies to aspirin, clopidogrel, or cilostazol thienopyridine use before enrollment
* concomitant use of other anti-thrombotic drugs (oral anticoagulants and dipyridamole)
* platelet count <100 x 106/μL
* hematocrit < 25%
* liver disease (bilirubin > 2 mg/dl)
* active bleeding or bleeding diathesis
* gastrointestinal bleeding within the last 6 months
* hemodynamic instability
* acute coronary or cerebrovascular event within 3 months
* malignancy
* concomitant use of a cytochrome P450 inhibitor or a non-steroidal anti-inflammatory drug
* recent treatment (<30 days) with a glycoprotein IIb/IIIa antagonist.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The differences of platelet aggregation according to the anti-platelet therapy. | 14 days
  Platelet function was assessed with light transmittance aggregometry and the VerifyNowTM P2Y12 assay.
  High on-treatment platelet reactivity was defined as 5 μmol/L of ADP-induced Aggmax > 50%.
  Inhibition of platelet aggregation (IPA) was defined as the percent decrease in aggregation values obtained at baseline and after treatment.
  VerifyNow-P2Y12 assay results are also assessed and expressed in P2Y12 reaction units (PRUs) and the percentage of inhibition.

SECONDARY OUTCOMES:
Changes of platelet activation markers according to the anti-platelet therapy | 14 days
  Markers of platelet activation (soluble CD40 ligand [sCD40L] and soluble P-selectin [sP-selectin]) were assessed at baseline and after 14 days of anti-platelet therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyunghee University
Locations (1):
- Kyung Hee University, Seoul, South Korea

REFERENCES:
- [Result] Park SH, Kim W, Park CS, Kang WY, Hwang SH, Kim W. A comparison of clopidogrel responsiveness in patients with versus without chronic renal failure. Am J Cardiol. 2009 Nov 1;104(9):1292-5. doi: 10.1016/j.amjcard.2009.06.049. PMID 19840579
- [Result] Angiolillo DJ, Shoemaker SB, Desai B, Yuan H, Charlton RK, Bernardo E, Zenni MM, Guzman LA, Bass TA, Costa MA. Randomized comparison of a high clopidogrel maintenance dose in patients with diabetes mellitus and coronary artery disease: results of the Optimizing Antiplatelet Therapy in Diabetes Mellitus (OPTIMUS) study. Circulation. 2007 Feb 13;115(6):708-16. doi: 10.1161/CIRCULATIONAHA.106.667741. Epub 2007 Jan 29. PMID 17261652
- [Result] Angiolillo DJ, Bernardo E, Capodanno D, Vivas D, Sabate M, Ferreiro JL, Ueno M, Jimenez-Quevedo P, Alfonso F, Bass TA, Macaya C, Fernandez-Ortiz A. Impact of chronic kidney disease on platelet function profiles in diabetes mellitus patients with coronary artery disease taking dual antiplatelet therapy. J Am Coll Cardiol. 2010 Mar 16;55(11):1139-46. doi: 10.1016/j.jacc.2009.10.043. PMID 20223369
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Woo JS, Kim W, Lee SR, Jung KH, Kim WS, Lew JH, Lee TW, Lim CK. Platelet reactivity in patients with chronic kidney disease receiving adjunctive cilostazol compared with a high-maintenance dose of clopidogrel: results of the effect of platelet inhibition according to clopidogrel dose in patients with chronic kidney disease (PIANO-2 CKD) randomized study. Am Heart J. 2011 Dec;162(6):1018-25. doi: 10.1016/j.ahj.2011.09.003. Epub 2011 Nov 8. PMID 22137075
- See also: Korea Food and Drug Administration — http://www.kfda.go.kr